CLINICAL TRIAL: NCT01511939
Title: Single Center, Open-label Study of Effect of PENNSAID (Diclofenac Sodium Solution Topical) on Coagulation Parameters (PT, PTT, INR and Platelet Function) in Patients With Moderate to Severe Osteoarthritis Pain of the Knee Taking Anticoagulant Medication
Brief Title: Trial to See if Topical Pennsaid for Knee Pain Affects Coagulation Values in Patients Who Are Also Taking Anticoagulants
Acronym: ATCCTCP-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nathan Wei, MD, FACP, FACR: (Other)
Collaborators: Medtronic - MITG (Industry); Arthritis Treatment Center, Maryland (Other)
Responsible Party: Sponsor-Investigator, Nathan Wei, MD, FACP, FACR:, Nathan Wei, MD, FACP, FACR, Arthritis Treatment Center, Maryland
Organization: Arthritis Treatment Center, Maryland (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ATCCTCP-1
Record Dates: First submitted 2012-01-09; First posted 2012-01-19 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Osteoarthritis of the Knee; Coagulopathy
Keywords: Knee pain; Anticoagulant; Warfarin; Dabigatran; Clopidogrel; Aspirin; Topical NSAID; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Hemostatic Disorders; Osteoarthritis | interventions — Diclofenac; Solutions; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pennsaid, warfarin (Other): Pennsaid 1.5%, 10 drops x 4 until 40 drops applied topically to index knee (and also non-index knee if osteoarthritis pain is present bilaterally) 4 times a day for a 4 week active treatment period in a subject who has been taking a stable dose of warfarin for at least 2 months
  Interventions: Drug: Pennsaid
- Pennsaid, dabigatran (Other): Pennsaid 1.5%, 10 drops x 4 until 40 drops applied topically to index knee (and also non-index knee if osteoarthritis pain is present bilaterally) 4 times a day for a 4 week active treatment period in a subject who has been taking a stable dose of dabigatran for at least 2 months
  Interventions: Drug: Pennsaid
- Pennsaid, aspirin and/or clopidogrel (Other): Pennsaid 1.5%, 10 drops x 4 until 40 drops applied topically to index knee (and also non-index knee if osteoarthritis pain is present bilaterally) 4 times a day for a 4 week active treatment period in a subject who has been taking a stable dose of aspirin and/or clopidogrel for at least 2 months
  Interventions: Drug: Pennsaid

INTERVENTIONS:
Drug: Pennsaid — Administered 10 drops x 4 until 40 drops applied topically to index knee (and also non-index knee if osteoarthritis pain is present bilaterally) 4 times a day for a 4 week active treatment period.
  Other Names: Pennsaid 1.5%; Diclofenac sodium 1.5% topical solution; Topical nonsteroidal antiinflammatory drug; Topical NSAID

SUMMARY:
The purpose of this study is to see if using a topical nonsteroidal antiinflammatory drug (Pennsaid) to treat osteoarthritis knee pain will affect coagulation values in patients who are also taking anticoagulant or antithrombotic medications.

DETAILED DESCRIPTION:
Open-label active treatment Phase III study of Pennsaid (diclofenac sodium 1.5% topical solution) to determine the effects on coagulation parameters in patients who are equal to or greater than 55 years of age with moderate to severe osteoarthritis knee pain and who are also taking warfarin, dabigatran, or aspirin and/or clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults > than or equal to 55
* Ambulatory subjects with moderate to severe osteoarthritis (OA) of the knee with symptoms and knee pain for at least 3 months and pain on the majority of days in the last 30 days.
* Subjects with bilateral knee OA, the more symptomatic knee is the index knee and PENNSAID can be applied on both knees if both are affected.
* Radiographic evidence of Kellgren-Lawrence Grade 2-4 within the past 2 years.
* Currently on a stable dose of anticoagulant therapy (warfarin, dabigatran, aspirin or clopidogrel) for the past 2 months and expected to remain on current dose for the six week duration of the study.
* If currently taking oral nonsteroidal antiinflammatory drug (NSAID) and/or acetaminophen for OA knee pain, must be taking it for at least an average of 25 days per month.
* Those currently taking oral NSAID must be willing to perform a 7 day washout to be eligible to be enrolled into the study.
* A pain score of > than 40mm on the Patient Pain Visual Analog Scale (VAS) (100 mm scale) at screening and baseline visit.
* Able to comply with the study and give informed consent prior to performance of any study procedures.
* Able to read, write and understand English.

Exclusion Criteria:

* Unwilling to abstain from oral NSAIDs and/or other analgesic medication except for acetaminophen as rescue medication. Subjects taking low dose aspirin for cardiovascular health may remain on their stable dose throughout the study.
* Unwilling to abstain from taking < than or equal to 1500mg of acetaminophen a day for rescue medication purposes during the 6 week course of the trial.
* Using a handicap assistance device i.e. cane, walker > than or equal to 50% of the time.
* Undergoing new physical therapy or participating in a weight loss or exercise program that has not been stable for at least 3 months prior to screening and won't remain stable during participation in study.
* History or diagnosis of an inflammatory arthritis i.e. rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, sarcoidosis, or amyloidosis.
* Known or clinically suspected infection and human immunodeficiency virus (HIV), or hepatitis C or B viruses.
* History of abnormal laboratory results > that or equal to 2.5 x upper limit of normal (ULN) indicative of any significant medical disease which in the opinion of the investigator, would preclude the subjects participation in the study.
* Any of the following abnormal laboratory results during screening:
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > than or equal to 2.5 x ULN
* Hemoglobin < than 11.5 g/dL (female) or < 13.2 g/dL (male)
* White blood cell count (WBC) < than 3500 cells/mm3
* Lymphocyte count < than or equal to 1000 cels/mm3
* Serum creatinine > than or equal 1.5 x ULN
* Platelet count below the central laboratory lower limit of normal (LLN)
* Coagulation tests (Prothrombin Time (PT), Partial Thromboplastin Time (PTT), International Normalized Ratio (INR), Platelet Aggregation) requiring an alteration in anticoagulant dosage.
* Skin breakdown or rash at knee where topical PENNSAID is to be applied.
* Other serious uncontrolled non-malignant, significant, acute or chronic medical or psychiatric illness that, in judgment of investigator, could compromise subject safety, limit subject's ability to complete study and/or compromise the objectives of study.
* History of malignancy in the past 5 years with exception of resected basal cell carcinoma, squamous cell carcinoma of the skin, or resected cervical atypia or carcinoma in situ.
* History of drug or alcohol dependence or abuse in the past 3 years.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Wei, MD,FACP,FACR, Principal Investigator — Arthritis Treatment Center, Frederick, Maryland, United States, 21702
Locations (1):
- Arthritis Treatment Center, Frederick, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pennsaid, Warfarin: Pennsaid 1.5%, 10 drops x 4 until 40 drops applied topically to index knee (and also non-index knee if osteoarthritis (OA) pain is present bilaterally) 4 times a day for a 4 week active treatment period in a subject who has been taking a stable dose of warfarin for at least 2 months
  Pennsaid: Administered 10 drops x 4 until 40 drops applied topically to index knee (and also non-index knee if OA pain is present bilaterally) 4 times a day for a 4 week active treatment period.
- Pennsaid, Dabigatran: Pennsaid 1.5%, 10 drops x 4 until 40 drops applied topically to index knee (and also non-index knee if OA pain is present bilaterally) 4 times a day for a 4 week active treatment period in a subject who has been taking a stable dose of dabigatran for at least 2 months
  Pennsaid: Administered 10 drops x 4 until 40 drops applied topically to index knee (and also non-index knee if OA pain is present bilaterally) 4 times a day for a 4 week active treatment period.
- Pennsaid, Aspirin and/or Clopidogrel: Pennsaid 1.5%, 10 drops x 4 until 40 drops applied topically to index knee (and also non-index knee if OA pain is present bilaterally) 4 times a day for a 4 week active treatment period in a subject who has been taking a stable dose of aspirin and/or clopidogrel for at least 2 months
  Pennsaid: Administered 10 drops x 4 until 40 drops applied topically to index knee (and also non-index knee if OA pain is present bilaterally) 4 times a day for a 4 week active treatment period.
Period: Overall Study
Arm/Group | Pennsaid, Warfarin | Pennsaid, Dabigatran | Pennsaid, Aspirin and/or Clopidogrel
Started | 9 (Includes 1 subject who was also taking aspirin.) | 5 (Includes one patient who was also taking aspirin.) | 8
Completed | 7 | 4 | 8
Not Completed | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: One subject in the warfarin group and one subject in the dabigatran group were also taking aspirin. For the Outcome measures, these two subjects were also included in the aspirin and/or clopidogrel group.
Groups:
- Pennsaid, Warfarin: Pennsaid 1.5%, 10 drops x 4 until 40 drops applied topically to index knee (and also non-index knee if OA pain is present bilaterally) 4 times a day for a 4 week active treatment period in a subject who has been taking a stable dose of warfarin for at least 2 months
  Pennsaid: Administered 10 drops x 4 until 40 drops applied topically to index knee (and also non-index knee if OA pain is present bilaterally) 4 times a day for a 4 week active treatment period.
- Total: Total of all reporting groups
Arm/Group | Pennsaid, Warfarin | Pennsaid, Dabigatran | Pennsaid, Aspirin and/or Clopidogrel | Total
Number analyzed (Participants) | 9 | 5 | 8 | 22
Age, Customized [Number; unit: participants]
  > / = 55 years | 9 | 5 | 8 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 5 | 15
  Male | 1 | 3 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 9 | 5 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in Laboratory Results of Prothrombin Time (PT)
Description: PT will be evaluated to determine if there is any significant effect of Pennsaid on coagulation parameters.
Time Frame: Baseline to week 4
Population: Two subjects who completed the study were taking both an anticoagulant medication and aspirin. For this analysis, the subject who was taking warfarin and aspirin was included only in the "Pennsaid, warfarin" group, and the subject who was taking dabigatran and aspirin was included only in the "Pennsaid, dabigatran" group.
Measure: Mean (Full Range); unit: seconds
Arm/Group | Pennsaid, Warfarin | Pennsaid, Dabigatran | Pennsaid, Aspirin and/or Clopidogrel
Number analyzed (Participants) | 7 | 4 | 8
seconds | 6.97 [0.20 to 10.80] | 0.96 [-2.40 to 2.30] | -0.04 [-0.80 to 0.70]

2. Primary Outcome: Change From Baseline to Week 4 in Laboratory Results of International Normalized Ratio (INR)
Description: INR will be evaluated to determine if there is any significant effect of Pennsaid on coagulation parameters.
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Mean (Full Range); unit: ratio
Arm/Group | Pennsaid, Warfarin | Pennsaid, Dabigatran | Pennsaid, Aspirin and/or Clopidogrel
Number analyzed (Participants) | 7 | 4 | 8
ratio | 0.63 [0.01 to 1.00] | 0.09 [-0.21 to 0.20] | 0.00 [-0.07 to 0.07]

3. Primary Outcome: Change From Baseline to Week 4 in Laboratory Results of Partial Thromboplastin Time (PTT)
Description: PTT will be evaluated to determine if there is any significant effect of Pennsaid on coagulation parameters.
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Mean (Full Range); unit: Seconds
Arm/Group | Pennsaid, Warfarin | Pennsaid, Dabigatran | Pennsaid, Aspirin and/or Clopidogrel
Number analyzed (Participants) | 7 | 4 | 8
Seconds | 2.68 [-1.20 to 6.30] | 1.50 [-5.80 to 7.20] | -0.29 [-2.90 to 2.30]

4. Primary Outcome: Change From Baseline to Week 4 in Laboratory Results of Platelet Aggregation
Description: Platelet Aggregation will be evaluated to determine if there is any significant effect of Pennsaid on coagulation parameters.
Time Frame: Baseline to Week 4
Population: For this analysis, the subject who was taking warfarin and aspirin was included in both the "Pennsaid, warfarin" group and the "Pennsaid, aspirin and/or clopidogrel" group, and the subject who was taking dabigatran and aspirin was included in both the "Pennsaid, dabigatran" group and the "Pennsaid, aspirin and/or clopidogrel" group.
Measure: Mean (Full Range); unit: Seconds
Arm/Group | Pennsaid, Warfarin | Pennsaid, Dabigatran | Pennsaid, Aspirin and/or Clopidogrel
Number analyzed (Participants) | 7 | 4 | 10
Seconds | 8.14 [-16.00 to 43.00] | -39.25 [-110.00 to -4.00] | -13.30 [-155.00 to 117.00]

ADVERSE EVENTS:
Arm/Group | Pennsaid, Warfarin | Pennsaid, Dabigatran | Pennsaid, Aspirin and/or Clopidogrel
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/5 | 0/10
Other Adverse Events (participants affected / at risk) | 6/9 | 0/5 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pennsaid, Warfarin (N=9) | Pennsaid, Dabigatran (N=5) | Pennsaid, Aspirin and/or Clopidogrel (N=10)
Epistaxis (General disorders) | 1 (1) | 0 (0) | 0 (0) — Epistaxis resulting in hospitalization and blood transfusion; assessed by Principal Investigator as not related to Pennsaid because patient had a history of sinus surgery which has resulted in a history of occasional severe epistaxis.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pennsaid, Warfarin (N=9) | Pennsaid, Dabigatran (N=5) | Pennsaid, Aspirin and/or Clopidogrel (N=10)
Bowel Impaction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Assessed by Principal Investigator as not related to Pennsaid
Swelling of lower extremities (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) — Assessed by Principal Investigator as possibly related to Pennsaid
Epistaxis (General disorders) | 1 (1) | 0 (0) | 0 (0) — Assessed by Principal Investigator as not related to Pennsaid
Broken Tooth (General disorders) | 1 (1) | 0 (0) | 0 (0) — Assessed by Principal Investigator as not related to Pennsaid
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) — Assessed by Principal Investigator as possibly related to Pennsaid
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Assessed by Principal Investigator as not likely related to Pennsaid
Rash on lower extremities (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Assessed by Principal Investigator as possibly related to Pennsaid
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) — Assessed by Principal Investigator as not related to Pennsaid
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Assessed by Principal Investigator as not related to Pennsaid
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Assessed by Principal Investigator as not related to Pennsaid
Metallic taste in mouth (General disorders) | 0 (0) | 0 (0) | 1 (1) — Assessed by Principal Investigator as possibly related to Pennsaid
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1) — Assessed by Principal Investigator as possibly related to Pennsaid
Hyperglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) — Assessed by Principal Investigator as not likely related to Pennsaid
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Assessed by Principal Investigator as not related to Pennsaid

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes